CLINICAL TRIAL: NCT02314247
Title: Multi-center, Phase 2, Open-label Study of Efficacy and Safety of the Selective Inhibitor of Nuclear Export (SINE™) Selinexor (KPT-330) in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL) and Cutaneous T-cell Lymphoma (CTCL)
Brief Title: Efficacy and Safety Study of Selinexor in Relapsed or Refractory Peripheral T-cell Lymphoma or Cutaneous T-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to enrollment challenges
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-013
Record Dates: First submitted 2014-12-03; First posted 2014-12-11 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Peripheral T-cell Lymphoma (PTCL); Cutaneous T-cell Lymphoma (CTCL)
Keywords: PTCL; CTCL; Peripheral T-cell Lymphoma; Cutaneous T-cell Lymphoma; Karyopharm; KPT-330; Selinexor
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selinexor (Experimental): 60 mg dose (equivalent to ~35 mg/m²)
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — 20 mg oral tablets: 60 mg dose on Days 1 and 3 of Weeks 1-4 of each 4-week cycle (Protocol V.3.0).
  20 mg oral tablets: 60 mg dose on Days 1 and 3 of Weeks 1-3 of each 4-week cycle (Protocol V.<3.0).
  Number of Cycles: up to 12 but there is no maximal duration for treatment.
  Other Names: KPT-330

SUMMARY:
This is a single-arm, multi-center, open-label phase 2 study of the SINE™ compound selinexor given orally to patients with relapsed or refractory PTCL or CTCL.

Approximately 60 patients with relapsed or refractory PTCL or CTCL who meet the eligibility criteria and have none of the exclusion criteria will be enrolled to receive selinexor until either disease progression or intolerance has occurred.

DETAILED DESCRIPTION:
This is a single-arm, multi-center, open-label phase 2 study of the SINE™ compound selinexor given orally to patients with relapsed or refractory PTCL or CTCL.

Approximately 60 patients with relapsed or refractory PTCL or CTCL who meet the eligibility criteria and have none of the exclusion criteria will be enrolled to receive selinexor until either disease progression or intolerance has occurred.

Enrolled patients will be given selinexor as an oral fixed 60 mg dose (equivalent to ~35 mg/m²) on Days 1 and 3 of Weeks 1-4 of each 4-week cycle (total 8 doses per cycle).

There is no maximum treatment duration. Patients will receive supportive therapy to mitigate selinexor side effects, as well as best supportive care (BSC).

Patients enrolled under Protocol Versions <3.0 were to receive selinexor orally, at a fixed dose of 60 mg (equivalent to ~35 mg/m²) on Days 1 and 3 of Weeks 1-3 of each 4-week cycle (total of 6 doses per cycle). Selinexor was not taken during Week 4.

For all patients enrolled in this study (regardless of the protocol version) who continued onto Cycle 3 and forward, the dose was to be increased by 20 mg to 80 mg (administered on Days 1 and 3 of Weeks 1-4), only after consultation with the Sponsor's Medical Monitor.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of ≤2.
* Relapsed or refractory disease to at least one prior systemic regimen.
* Measurable disease: according to International Working Group (IWG) guidelines for all patients with PTCL and according to CTCL Response in Skin consensus criteria for all patients with CTCL.
* Objective, documented evidence of disease progression on study entry.

Exclusion Criteria:

* Known active central nervous system (CNS) lymphoma.
* Active graft-versus-host disease after allogeneic stem cell transplantation. At least 4 months must have elapsed since completion of allogeneic stem cell transplantation.
* Unable to swallow tablets or malabsorption syndrome, disease significantly affecting gastrointestinal function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (4):
  - Concord Repatriation General Hospital (CRGH), Concord, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Cabrini Hospital, Malvern, Victoria
- National Cancer Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Selinexor (PTCL); Selinexor (CTCL): Assigned to 60 mg dose twice weekly
- Selinexor (CTCL) 8 Doses/Cycle: Assigned to 60 mg dose twice weekly for weeks 1-4
Period: Overall Study
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL) | Selinexor (CTCL) 8 Doses/Cycle
Started | 9 | 6 | 1
Completed | 0 | 0 | 0
Not Completed | 9 | 6 | 1
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 1
Not completed — Progression of Disease | 6 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Selinexor (PTCL): Assigned to 60 mg dose, 6 doses/cycle
- Selinexor (CTCL): Assigned to 60 mg dose, 6 doses/cycle (6 patients); Assigned to 60 mg dose, 8 doses/cycle (1 patient)
- Total: Total of all reporting groups
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL) | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Median (Full Range); unit: years] | 65 [51 to 83] | 74 [59 to 84] | 69 [51 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall Response (OR) = Complete Response (CR) + Partial Response (PR). Objective disease response assessment in PTCL patients was made according to the revised response criteria based on the International Working Group (IWG) guidelines for malignant lymphoma (Cheson, 2007). Objective disease response assessment in CTCL patients was assessed according to the revised CTCL Consensus Response Criteria (Olsen, 2011) using physical examination, including the Modified Severity Weighted Assessment Tool (mSWAT) for skin assessment. CTCL Global Response Score was used as a secondary efficacy assessment. Progression was defined as the first occurrence of progressive disease (PD) per the revised response criteria. Clinical disease progression in the absence of formal criteria for PD must be documented by a physician.
Time Frame: Disease response was assessed at screening and every 8 weeks (patients with PTCL); or at Cycle 1 Day 1 and every 4 weeks (patients with CTCL), until disease progression.
Population: Due to the limited enrollment in this study, only the Intent to Treat (ITT) Population, consisting of all patients who received at least 1 dose of study treatment (which is identical to the Safety Population), was evaluated for efficacy.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
Number analyzed (Participants) | 9 | 7
Percentage of participants | 11.1 [1.2 to 36.8] | 14.3 [1.5 to 45.3]

2. Primary Outcome: Best Overall Response: Complete Response (CR)
Description: Patients who achieved CR (disappearance of all detectable evidence of disease). Objective disease response assessment in PTCL patients was made according to the revised response criteria based on the International Working Group (IWG) guidelines for malignant lymphoma (Cheson, 2007). Objective disease response assessment in CTCL patients was assessed according to the revised CTCL Consensus Response Criteria (Olsen, 2011) using physical examination, including the Modified Severity Weighted Assessment Tool (mSWAT) for skin assessment. CTCL Global Response Score was used as a secondary efficacy assessment.
Time Frame: as for outcome 1
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

3. Primary Outcome: Best Overall Response: Partial Response (PR)
Description: Patients whose best overall response to study treatment was PR (regression of measurable disease and no new sites). Objective disease response assessment in PTCL patients was made according to the revised response criteria based on the International Working Group (IWG) guidelines for malignant lymphoma (Cheson, 2007). Objective disease response assessment in CTCL patients was assessed according to the revised CTCL Consensus Response Criteria (Olsen, 2011) using physical examination, including the Modified Severity Weighted Assessment Tool (mSWAT) for skin assessment. CTCL Global Response Score was used as a secondary efficacy assessment.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) population
Measure: Count of Participants; unit: Participants
Groups:
- Selinexor (PTCL): Assigned to 60 mg dose; 6 doses/cycle
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
Number analyzed (Participants) | 9 | 7
Participants | 1 | 1

4. Primary Outcome: Best Overall Response: Stable Disease (SD)
Description: Patients whose best overall response to study treatment was SD (failure to attain criteria needed for CR or PR, or to meet criteria for PD). Objective disease response assessment in PTCL patients was made according to the revised response criteria based on the International Working Group (IWG) guidelines for malignant lymphoma (Cheson, 2007). Objective disease response assessment in CTCL patients was assessed according to the revised CTCL Consensus Response Criteria (Olsen, 2011) using physical examination, including the Modified Severity Weighted Assessment Tool (mSWAT) for skin assessment. CTCL Global Response Score was used as a secondary efficacy assessment.
Time Frame: as for outcome 1
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
Number analyzed (Participants) | 9 | 7
Participants | 2 | 4

5. Primary Outcome: Best Overall Response: Progressive Disease (PD)
Description: Patients whose best overall response to study treatment was PD. Progression was defined as the first occurrence of progressive disease (PD). Objective disease response assessment in PTCL patients was made according to the revised response criteria based on the International Working Group (IWG) guidelines for malignant lymphoma (Cheson, 2007). Objective disease response assessment in CTCL patients was assessed according to the revised CTCL Consensus Response Criteria (Olsen, 2011) using physical examination, including the Modified Severity Weighted Assessment Tool (mSWAT) for skin assessment. CTCL Global Response Score was used as a secondary efficacy assessment. Clinical disease progression in the absence of formal criteria for PD must be documented by a physician.
Time Frame: as for outcome 1
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
Number analyzed (Participants) | 9 | 7
Participants | 2 | 0

6. Primary Outcome: Best Overall Response: Not Evaluable (NE)
Description: Patients who could not be assessed quantitatively for disease response for any reason.
Time Frame: as for outcome 1
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
Number analyzed (Participants) | 9 | 7
Participants | 4 | 2

7. Secondary Outcome: Duration of Stable Disease, Including Patients With Partial Response
Description: Duration of time from the date of start of study treatment to the date of disease progression. Objective disease response assessment in PTCL patients was made according to the revised response criteria based on the International Working Group (IWG) guidelines for malignant lymphoma (Cheson, 2007). Objective disease response assessment in CTCL patients was assessed according to the revised CTCL Consensus Response Criteria (Olsen, 2011) using physical examination, including the Modified Severity Weighted Assessment Tool (mSWAT) for skin assessment. CTCL Global Response Score was used as a secondary efficacy assessment.
Time Frame: Date of start of study treatment to date of progression. Patients without documented PD are censored on date of last radiologic assessment.
Population: Those participants with stable disease, including those with partial response, as a subset of the Intent to Treat (ITT) population
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Selinexor (PTCL); Selinexor (CTCL): Assigned to 60 mg, 6 doses/cycle
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
Number analyzed (Participants) | 3 | 5
Days | 120.5 [111.0 to 130.0] | 112.0 [85.0 to 225.0]

8. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of patients who have CR, PR, or SD lasting ≥ 8 weeks. Objective disease response assessment in PTCL patients was made according to the revised response criteria based on the International Working Group (IWG) guidelines for malignant lymphoma (Cheson, 2007). Objective disease response assessment in CTCL patients was assessed according to the revised CTCL Consensus Response Criteria (Olsen, 2011) using physical examination, including the Modified Severity Weighted Assessment Tool (mSWAT) for skin assessment. CTCL Global Response Score was used as a secondary efficacy assessment.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) Population
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
Number analyzed (Participants) | 9 | 7
Percentage of participants | 33.3 [12.9 to 59.9] | 71.4 [40.4 to 92.1]

9. Secondary Outcome: Progression Free Survival (PFS)
Description: Duration of time from start of study treatment to date of disease progression or death from any cause.
Time Frame: Study treatment start date to date of disease progression or date of death. Patients without documented PD are censored on date of last radiologic assessment.
Population: Intent to Treat population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
Number analyzed (Participants) | 9 | 7
Days | 111.0 [41.0 to 130.0] | 112.0 [85.0 to 225.0]

ADVERSE EVENTS:
Time Frame: Day of onset after the first dose of study treatment through 30 days following the last dose of study treatment.
Description: All patients who received at least 1 dose of study treatment were included in the Safety Population.
Groups:
- Selinexor (PTCL): Assigned to 60 mg; 6 doses/cycle
- Selinexor (CTCL): Assigned to 60 mg; 6 doses/cycle (6 patients)
  Assigned to 60 mg; 8 doses/cycle (1 patient)
Arm/Group | Selinexor (PTCL) | Selinexor (CTCL)
All-Cause Mortality (participants affected / at risk) | 3/9 | 1/7
Serious Adverse Events (participants affected / at risk) | 8/9 | 1/7
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selinexor (PTCL) (N=9) | Selinexor (CTCL) (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selinexor (PTCL) (N=9) | Selinexor (CTCL) (N=7)
Nausea (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 1 | 4
Diarrhea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 5
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0
Vision Blurred (Eye disorders) | 2 | 1
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1
Mean Cell Haemoglobin Concentration Increased (Investigations) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue (General disorders) | 4 | 5
Pyrexia (General disorders) | 1 | 0
Feeling Cold (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Peripheral Swelling (General disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Amnesia (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to unexpectedly slow recruitment, the Sponsor decided to terminate the study after 16 patients had been enrolled. The small study population limits the evaluation of both efficacy and safety of selinexor in patients with PTCL or CTCL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes